CLINICAL TRIAL: NCT05715905
Title: An In Depth Study Evaluating Patterns in the Colon Cancer Patients Clinical Trials
Brief Title: Analyzing Clinical Trial Experiences of Colon Cancer Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 81122503
Record Dates: First submitted 2023-01-27; First posted 2023-02-08 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Colon Cancer; Colon Disease
Keywords: Colon Cancer; Colon Disease
MeSH Terms: conditions — Colonic Neoplasms; Colonic Diseases

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Participation in medical trials usually favors a particular demographic group. But there is limited research available to explain what trial attributes affect the completion of these specific demographic groups.

This trial will admit a wide range of data on the clinical trial experience of Colon Cancer patients to determine which factors prevail in limiting a patient's ability to join or finish a trial.

It will also try to analyze data from the perspective of different demographic groups to check for recurring trends which might yield insights for the sake of future Colon Cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been diagnosed with colon cancer
* Patient has self-identified as planning to enroll in an observational clinical trial
* Patient is a minimum of 18 years or older

Exclusion Criteria:

* Pregnant or nursing patients
* Inability to perform regular electronic reporting
* Patient does not understand, sign, and return consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Colon cancer patients who are actively considering participating in a clinical trial, but have not yet completed enrollment and randomization.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Number of colon cancer patients who decide to enroll in a clinical trial | 3 months
Rate of patients who remain in a colon cancer clinical trial to trial completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Labianca R, Beretta GD, Kildani B, Milesi L, Merlin F, Mosconi S, Pessi MA, Prochilo T, Quadri A, Gatta G, de Braud F, Wils J. Colon cancer. Crit Rev Oncol Hematol. 2010 May;74(2):106-33. doi: 10.1016/j.critrevonc.2010.01.010. PMID 20138539
- [Background] Mody K, Bekaii-Saab T. Clinical Trials and Progress in Metastatic Colon Cancer. Surg Oncol Clin N Am. 2018 Apr;27(2):349-365. doi: 10.1016/j.soc.2017.11.008. PMID 29496094
- [Background] Iqbal A, George TJ. Randomized Clinical Trials in Colon and Rectal Cancer. Surg Oncol Clin N Am. 2017 Oct;26(4):689-704. doi: 10.1016/j.soc.2017.05.008. Epub 2017 Aug 18. PMID 28923225

DOCUMENTS (1):
  • Informed Consent Form (2023-01-27): https://cdn.clinicaltrials.gov/large-docs/05/NCT05715905/ICF_000.pdf